CLINICAL TRIAL: NCT00553800
Title: Phase II Study of Bevacizumab and Erlotinib in Elderly Patients With Advanced Non-Small Lung Cancer
Brief Title: Study of Bevacizumab and Erlotinib in Patients With Advanced Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-TH-007
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab & Erlotinib (Experimental): bevacizumab 15 mg/kg intravenous every three weeks and erlotinib pill 150 mg by mouth every day
  Interventions: Drug: bevacizumab; Drug: Erlotinib

INTERVENTIONS:
Drug: bevacizumab
  Other Names: Other names: Avastin
Drug: Erlotinib
  Other Names: Other name: Tarceva

SUMMARY:
This study will evaluate the combination of bevacizumab and erlotinib in elderly patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
There is no definite evidence of a superior therapy for advanced non-small cell lung cancer in elderly patients. With the exception of one known study, single agent erlotinib has not been studied exclusively in the elderly and the combination of erlotinib and bevacizumab has never been studied exclusively in the treatment naive elderly. This is an important population that needs less toxic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologic confirmed non-small cell lung cancer, stage IIIB or IV or recurrent after primary surgery or radiotherapy.
* ECOG PS 0-1
* 70 years of age or older
* Must have measurable disease
* ANC > 1500, platelets > 100,000
* Total bilirubin </= 1.5, SGOT * SGPT < 5 x ULN
* Able and willing to swallow and absorb oral medication
* Able and willing to sign consent
* Request archival diagnostic tissue for EGFR expression but not required

Exclusion Criteria:

* Proteinuria as demonstrated by UPC ratio >/= 1.0
* Prior treatment with an investigational or marketed inhibitor of the EGFR pathway or anti-angiogenesis agent (includes thalidomide)
* Prior treatment for advanced stage disease, with the exception of surgery or radiation (no systemic)
* History of gross hemoptysis within 1 month of enrollment unless treated with surgery or radiation
* Evidence of bleeding diathesis or coagulopathy or other serious/acute internal bleeding within 6 months of enrollment.
* Current, ongoing treatment with full dose warfarin or equivalent
* Current(within 10 days)use of aspirin (> 325mg/day) or other NSAID with antiplatelet activity
* History of hemorrhagic or thrombotic stoke, TIA, or other CNS bleeding w/in last 6 months. Clinically significant PVD
* Known CNS disease except for treated brain mets.
* Squamous cell histology
* Blood pressure > 150/100 that cannot be ameliorated with standard anti-hypertensives
* History of hypertensive crisis or hypertensive encephalopathy
* NYHA grade II or > CHF
* History of MI within 6 months of enrollment
* Major surgery, open biopsy, significant trauma within 28 days of enrollment
* Pregnancy, lactation
* Abdominal or other fistula, abcess, perforation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2011-01-12 (Actual); Study Completion 2011-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Borghaei, DO, Principal Investigator — Fox Chase Cancer Center
Locations (7):
- United States (7):
  - AtlantiCare Regional Medical Center, Galloway, New Jersey
  - Fox Chase Virtua Health Cancer Program at Memorial, Mount Holly, New Jersey
  - Paoli Hospital, Paoli, Pennsylvania
  - Abramson Cnacer Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phase II study of bevacizumab and erlotinib in treatment-naïve elderly patients (older than age 65) with advanced non-small cell lung cancer (NSCLC). H. Borghaei, R. Mehra, M. M. Millenson, H. Tuttle, K. Ruth, A. J. Magdalinski, D. M. Mintzer, J. W. Lee, G. R. Simon, and C. J. Langer Journal of Clinical Oncology 2010 28:15_suppl, e18019-e18019

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab & Erlotinib: bevacizumab 15 mg/kg intravenous every three weeks and erlotinib pill 150 mg by mouth every day
  bevacizumab
  Erlotinib
Period: Overall Study
Arm/Group | Bevacizumab & Erlotinib
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab & Erlotinib
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  ≤ 75 yrs | 18
  > 75 yrs | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 26
  African-American | 5
  Native American | 1
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab & Erlotinib
Number analyzed (Participants) | 32
months | 6.6 [3.2 to 12.0]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Bevacizumab & Erlotinib
All-Cause Mortality (participants affected / at risk) | 17/32
Serious Adverse Events (participants affected / at risk) | 15/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab & Erlotinib (N=32)
Dehydration (Metabolism and nutrition disorders) | 3
FTT (Metabolism and nutrition disorders) | 1
Pain (General disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Anemia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 2
Fatigue (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2
Bowel perforation (Gastrointestinal disorders) | 1
Hypoxia (Cardiac disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab & Erlotinib (N=32)
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 10
Anorexia (Gastrointestinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 13
Nail changes (Skin and subcutaneous tissue disorders) | 3
Dry cracked skin (Skin and subcutaneous tissue disorders) | 8
Fissures (Skin and subcutaneous tissue disorders) | 2
Incr. hair growth (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Fatigue (General disorders) | 10
Weight loss (Metabolism and nutrition disorders) | 7
Depression (Psychiatric disorders) | 7
Neuropathy (Nervous system disorders) | 7
Hypertension (Vascular disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Deep vein thrmbosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT00553800/Prot_SAP_000.pdf